CLINICAL TRIAL: NCT04503707
Title: French Prospective Multicentre Non-Interventional Study to Assess the Design of Use of REKOVELLE® in Women Undergoing In Vitro Fertilisation or Intracytoplasmic Sperm Injection Procedures in Routine Clinical Practice
Brief Title: Study to Assess the Design of Use of REKOVELLE® in Women Undergoing In Vitro Fertilisation or Intracytoplasmic Sperm Injection Procedures in Routine Clinical Practice
Acronym: DELTA
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000370
Record Dates: First submitted 2020-06-26; First posted 2020-08-07 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Controlled Ovarian Stimulation
Keywords: Follicle Stimulating Hormone (FSH); Assisted Reproductive Technologies (ART); Follitropin Delta; REKOVELLE
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follitropin Delta: Treatment according to routine clinical practice.
  Interventions: Drug: Follitropin Delta

INTERVENTIONS:
Drug: Follitropin Delta — The Intervention (solution for injection) is delivered with a pre-filled injection pen. The REKOVELLE dose will be based on a recent determination (within the last 12 months) of AMH (anti- müllerian hormone) measured by the ELECSYS AMH Plus Immunoassay.
  Other Names: REKOVELLE

SUMMARY:
The aim of the study is to explore how the individualized dosing regimen of REKOVELLE is used in routine clinical practice and to describe the effectiveness and safety of REKOVELLE under real-world conditions.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older at enrolment
* Who are treated for IVF or ICSI treatment cycle using fresh or frozen ejaculated sperm from male partner or sperm donor
* Who are prescribed REKOVELLE for the first time and using the dosing algorithm to define the dose regimen: a previous cycle with REKOVELLE should not be allowed
* Who have been informed verbally and in writing about this study content and who do not object to their data being electronically processed.

Exclusion Criteria:

* Participating in an interventional clinical trial in which any treatment or follow-up is mandated
* Women with a contraindication for prescription of REKOVELLE treatment
* Oocyte donors
* Women undergoing ovarian stimulation for fertility preservation
* Women undergoing their third or fourth attempt of IVF or ICSI for the current parental project.
* Subject non-affiliated to French Social Security
* Women placed under judicial protection, guardianship, or supervision

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who are prescribed REKOVELLE within the approved indication for in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatment will be invited to participate in the study. Subjects will be enrolled only after the treatment decision has been made and no aspect of this study will interfere with or influence the routine medical procedures and/or medications received.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Daily dose of REKOVELLE administered (for naïve and non-naïve subjects) | At the end of the stimulation protocol (up to 30 days)
Duration of treatment with REKOVELLE (for naïve and non-naïve subjects) | From first until last day of REKOVELLE treatment (up to 30 days)
Use of the dosing App (for naïve and non-naïve subjects) | At visit when the daily dose of REKOVELLE is decided (up to 2 hours)
Type of Gonadotropin-Releasing Hormone (GnRH) used (for naïve and non-naïve subjects) | At visit (up to 2 hours) during the REKOVELLE treatment period
Duration of treatment with GnRH (for naïve and non-naïve subjects) | At the end of the ovarian controlled stimulation (up to 2 weeks)
Treatment used for the triggering of follicle maturation (for naïve and non-naïve subjects) | At the last visit during the REKOVELLE treatment period (from 5 to 30 days)
Treatment used for Luteal phase support (for naïve and non-naïve subjects) | From start of REKOVELLE treatment until 10-11 weeks after embryo transfer
  Decided as a choice between Progesterone, Oestrogen and hCG

SECONDARY OUTCOMES:
Rate of Ongoing Pregnancy (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Ongoing pregnancy is defined as at least one intrauterine viable fetus, 10-11 weeks after first fresh or frozen embryo/blastocyst transfer.
Number of oocytes retrieved (for naïve and non-naïve subjects) | At visit (up to 2 hours) at 36 hours after completed REKOVELLE treatment
Number of oocytes/embryos/blastocysts frozen (for naïve and non-naïve subjects) | At Day 3 after oocyte retrieval
Quality of fresh or frozen embryos or blastocysts transferred (excellent, good, fair, other) (for naïve and non-naïve subjects) | At Day 3, 5 or 6 after oocyte retrieval
Implantation rate (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Implantation rate is defined as number of intrauterine viable fetus after transfer divided by the number of embryos/blastocysts transferred.
Positive human chorionic gonadotropin (hCG) test (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Proportion of subjects with positive hCG test.
Clinical pregnancy rate (for naïve and non-naïve subjects) | Up to 5-6 weeks after transfer
  Clinical pregnancy is defined as least one gestational sac.
Incidence of biochemical pregnancy (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Biochemical pregnancy is defined as positive beta hCG (βhCG) test but no gestational sac is observed on later transvaginal ultrasound, or menstruation is reported.
Incidence of spontaneous abortion (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Spontaneous abortion is defined as positive βhCG test but all intrauterine gestational sacs without fetal heart beat as documented by ultrasound, or there are no viable fetuses observed by ultrasound.
Incidence of elective abortion (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Elective abortion is defined as induced abortion done at the request of the woman for other than therapeutic reasons.
Incidence of vanishing twins (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Vanishing twin is defined as spontaneous disappearance of an intrauterine gestational sac with or without heart beat in a pregnancy where one viable fetus remains as documented by ultrasound.
Incidence of ectopic pregnancy (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Ectopic pregnancy is defined as extrauterine gestational sac with or without fetal heart beat as documented by ultrasound or surgery.
Proportion of subjects with cycle cancellation (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Cancellation could be done before oocyte pick up (due to poor ovarian response, excessive ovarian response, any illness which prevents oocyte collection procedure, subject not taking hCG injection at the correct time, subject choice, other) or after oocyte pick up (due to no oocytes collected, no oocytes fertilized, abnormal fertilization, abnormal embryo development, no embryo development, ovarian hyperstimulation syndrome (OHSS), subject choice, other)
Type of gonadotropin used (previous cycle information for non-naïve subjects) | At baseline
Dose of gonadotropin used (previous cycle information for non-naïve subjects) | At baseline
Duration of treatment with gonadotropin (previous cycle information for non-naïve subjects) | At baseline
Type of GnRH used (previous cycle information for non-naïve subjects) | At baseline
  Defined as a choice between GnRH agonist and GnRH antagonist
Duration of treatment with GnRH (previous cycle information for non-naïve subjects) | At baseline
Treatment used for the triggering of follicle maturation (previous cycle information for non-naïve subjects) | At baseline
Treatment used for Luteal phase support (previous cycle information for non-naïve subjects) | At baseline
  Decided as a choice between Progesterone, Oestrogen and hCG
Number of oocytes retrieved (previous cycle information for non-naïve subjects) | At baseline
Number of embryos/blastocysts transferred (previous cycle information for non-naïve subjects) | At baseline
Incidence of pregnancy loss in women with embryo/blastocyst transfer (previous cycle information for non-naïve subjects) | At baseline
  Pregnancy loss included biochemical pregnancy, spontaneous / elective abortion, ectopic pregnancy.
Proportion of subjects with OHSS including moderate/severe grade (previous cycle information for non-naïve subjects) | At baseline
  Each OHSS case will be classified as moderate or severe.
Proportion of subjects with preventive interventions for early OHSS (previous cycle information for non-naïve subjects) | At baseline
  Preventive interventions cover triggering of final follicular maturation with GnRH agonist and fresh embryo/blastocyst transfer or cryopreservation of oocytes/embryos/blastocysts, cycle cancellation, coasting.
Proportion of subjects with preventive interventions for early OHSS (for naïve and non-naïve subjects) | Up to 10-11 weeks after transfer
  Preventive interventions cover triggering of final follicular maturation with GnRH agonist and fresh embryo/blastocyst transfer or cryopreservation of oocytes/embryos/blastocysts, Cycle cancellation, Coasting.
Frequency of adverse drug reactions (ADR) (for naïve and non-naïve subjects) | From start of REKOVELLE treatment until 10-11 weeks after embryo transfer
  An ADR is characterized by the causal relationship between REKOVELLE and the adverse event is at least a reasonable possibility.
Monitoring of the REKOVELLE treatment (number and intents of each visit) (for naïve and non-naïve subjects) | From Day 1 up to the last day of REKOVELLE stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (14):
- France (14):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Hopital Antoine Béclère, Clamart
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre hospitalier de Lille-Hopital de Flandre, Lille
  - Institut de Médecine de la Reproduction (there may be other sites in this country), Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes Hôpital Hôtel Dieu, Nantes
  - Maternité Port Royal, Paris
  - Centre Hospitalier Intercommunal de Poissy, Poissy
  - Clinique Mutualiste La Sagesse, Rennes
  - Pierre OGER, Rueil-Malmaison
  - CMCO, Strasbourg
  - CHU Toulouse - Hôpital Paule de Viguier, Toulouse